CLINICAL TRIAL: NCT06017895
Title: Doxepin Solution for Alleviation of Stubborn Breakthrough Pain Induced by Swallowing in Patient Receiving Radiotherapy for Nasopharyngeal Carcinoma: A Multicenter, Randomized, Controlled, Double-Blind Clinical Trial
Brief Title: Doxepin Solution for Alleviation of Stubborn Breakthrough Pain Induced by Swallowing in Patients Receiving Radiotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NFEC-2023-351
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Swallowing-induced Pain
Keywords: Nasopharyngeal carcinoma; Oral mucositis; Radiotherapy; Swallowing-induced pain; Doxepin
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Stomatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doxepin solution (Experimental): Patients received a doxepin solution spray to the posterior pharyngeal wall 10 minutes before eating. At least 12 hours later, when the swallowing-induced pain score ≥4, a placebo spray was administered to the posterior pharyngeal wall 10 minutes before eating.
  Interventions: Drug: doxepin solution
- placebo (Placebo Comparator): Patients received a placebo spray to the posterior pharyngeal wall 10 minutes before eating. At least 12 hours later, when the swallowing-induced pain score ≥4, a doxepin solution spray was administered to the posterior pharyngeal wall 10 minutes before eating.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: doxepin solution — 2.0 mL doxepin solution (5mg/mL) sprayed to the posterior pharyngeal wall
  Arms: doxepin solution
Other: Placebo — 2.0 mL placebo sprayed to the posterior pharyngeal wall
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to explore the effectiveness and adverse reactions of doxepin solution spray for alleviation of stubborn breakthrough pain induced by swallowing in patients receiving radiotherapy for nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Patients with nasopharyngeal carcinoma receiving radical radiotherapy or chemoradiotherapy who developed oral mucositis and had a swallowing-induced pain score ≥ 4 were recruited and randomly assigned 1:1 to the experimental group and the control group.

Patients in the experimental group received a doxepin solution spray to the posterior pharyngeal wall 10 minutes before eating. At least 12 hours later, when the swallowing-induced pain score ≥4, a placebo spray was administered to the posterior pharyngeal wall 10 minutes before eating.

Patients in the control group received a placebo spray to the posterior pharyngeal wall 10 minutes before eating. At least 12 hours later, when the swallowing-induced pain score ≥4, a doxepin solution spray was administered to the posterior pharyngeal wall 10 minutes before eating.

The swallowing-induced pain and incidence of adverse events were assessed at 10 minutes, 20 minutes, 30 minutes, and 1 hour after medication using a patient-reported questionnaire, and safety evaluation was conducted 1 day after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed written consent.
2. Age ≥ 18 years.
3. Histologically confirmed as nasopharyngeal carcinoma, and currently undergoing radical radiotherapy or chemoradiotherapy.
4. Physical examination demonstrating the presence of radiation-induced mucositis in the oral cavity and/or oropharynx.
5. At least 4 (out of 10) patient-reported swallowing-induced pain as measured by the numeric rating scale of pain.
6. Being able to complete the questionnaires independently or with assistance.
7. ECOG Performance Status 0, 1 or 2.

Exclusion Criteria:

1. Known allergy to doxepin, tricyclic antidepressants, or any known component of the drug formulation.
2. Use of a tricyclic antidepressant or monoamine oxidase inhibitor within 14 days prior to registration.
3. Current untreated or unhealed oral candidiasis or oral herpes simplex virus infection.
4. Untreated narrow angle glaucoma within 6 weeks prior to registration.
5. Untreated urinary retention within 6 weeks prior to registration.
6. Administration of cryotherapy to prevent oral mucositis within 6 weeks prior to registration.
7. Current serious heart disease or a recent history of myocardial infarction.
8. Current untreated or unresolved conditions like epilepsy, hyperthyroidism, hepatic dysfunction, delirium, and neutropenia.
9. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Redution of swallowing-induced pain | Baseline, and 10, 20, 30, 60 minutes after administration
  The redution of swallowing-induced pain was measured by the numerical analogue scale of 0 to 10, with 0=no pain and 10=worst pain in the questionnaires taken at baseline, and 10, 20, 30, 60 minutes after assigned administration.

SECONDARY OUTCOMES:
Total Drowsiness Increase | Baseline, and 10, 20, 30, 60 minutes after administration
  The total drowsiness increase was measured by the numerical analogue scale of 0 to 10, with 0=no drowsiness and 10=extreme drowsiness in the questionnaires taken at baseline, and 10, 20, 30, 60 minutes after assigned administration.
Total Taste of the Agent | 10, 20, 30 and 60 minutes after administration
  The total taste of the agent was measured by the numerical analogue scale of 0 to 10, with 0=acceptable and 10=terrible in the questionnaires taken at 10, 20, 30 and 60 minutes after assigned administration.
Total Stinging or Burning From the Agent | 10, 20, 30 and 60 minutes after administration
  The stinging or burning of the oral cavity/oropharynx was measured by the numerical analogue scale of 0 to 10, with 0=no stinging or burning and 10=worst stinging or burning in the questionnaires taken at 10, 20, 30 and 60 minutes after assigned administration.
Difficulty in Swallowing Different Food | Baseline, and 10, 20, 30, 60 minutes after administration
  The difficulty in swallowing liquids, pureed food and solid food was measured respectively by the numerical analogue scale of 0 to 10, with 0=not at all and 10=very much in the questionnaires taken at 10, 20, 30 and 60 minutes after assigned administration.
Patient Preference for Continuing Therapy With the Agent | 60 minutes after administration
  Patients were asked if they would like to continue treatment with that particular agent at 60 minutes after assigned administration.
Adverse Event Profiles | up to one day after administration
  Adverse events were assessed and record using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Guan, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Southern medical university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No